CLINICAL TRIAL: NCT02296554
Title: SLAP Repair Versus Biceps Tenodesis for SLAP Tears in the Shoulder: A Randomized Outcomes Study
Brief Title: Superior Labral Tear From Anterior to Posterior (SLAP) Repair Versus Biceps Tenodesis for SLAP Tears in the Shoulder
Acronym: SLAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: HealthPartners Institute (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1401M47421
Record Dates: First submitted 2014-11-10; First posted 2014-11-20 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2018-11

CONDITIONS: SLAP Tear
Keywords: SLAP Repair; Biceps Tenodesis
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLAP Repair (Experimental): Patient will receive SLAP repair for their SLAP tear.
  Interventions: Procedure: SLAP Repair
- Biceps Tenodesis Repair (Experimental): Patient will receive biceps tenodesis repair for their SLAP tear.
  Interventions: Procedure: Biceps Tenodesis

INTERVENTIONS:
Procedure: SLAP Repair — SLAP repair for SLAP tear
  Arms: SLAP Repair
Procedure: Biceps Tenodesis — Biceps tenodesis for SLAP tear
  Arms: Biceps Tenodesis Repair

SUMMARY:
Biceps Tenodesis is currently advocated for older, less active patients, but to date is not often advocated for Superior Labral Tear from Anterior to Posterior (SLAP) tears in young, active patients. The ideal surgical management for this pathology is not clearly known. More surgeons are using biceps tenodesis as a treatment for SLAP tears, including in the young, active population. If this study were to demonstrate that biceps tenodesis is similar to or better than SLAP repair, this would fundamentally change the treatment of SLAP tears. Perhaps more importantly, it would likely mean a less involved rehabilitation and earlier return to activities for patients with this pathology.

ELIGIBILITY:
Inclusion Criteria:

- Primary isolated SLAP tear, confirmed on MRI

Exclusion Criteria:

* Concomitant procedure needed such as a labral repair, rotator cuff repair or distal clavicle excision.
* Revision Surgery
* Previous shoulder surgery
* Major medical illness
* Inability to speak or read English

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Patient reported function and pain | Baseline
  American Shoulder and Elbow Surgeons (ASES)
Patient reported function and pain | 6 months
  ASES
Patient reported function and pain | 1 year
  ASES
Patient reported function and pain | 2 years
  ASES
Patient reported function and pain | 5 years
  ASES

SECONDARY OUTCOMES:
Range of Motion & Strength | Baseline
  Shoulder/elbow range of motion and strength measurements
Range of Motion | 3 months
  Shoulder/elbow range of motion
Range of Motion & Strength | 6 months
  Shoulder/elbow range of motion and strength measurements
Range of Motion & Strength | 1 year
  Shoulder/elbow range of motion and strength measurements
Range of Motion & Strength | 2 years
  Shoulder/elbow range of motion and strength measurements

CONTACTS AND LOCATIONS:
Locations (1):
- TRIA Orthopaedic Center, Bloomington, Minnesota, United States